CLINICAL TRIAL: NCT02646917
Title: A Single-Center Trial to Evaluate the Efficacy and Tolerability of SkinPen on Male and Female Subjects' Acne Scars on the Face and/or Back
Brief Title: SkinPen Efficacy on Acne Scars on the Face and/or Back
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bellus Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bellmed001
Record Dates: First submitted 2015-12-21; First posted 2016-01-06 (Estimated); Results first posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Atrophic Acne Scar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SkinPen II (Active Comparator): Three treatments using SkinPen II aesthetic microneedling device to each patient, with each treatment spaced one month apart.
  Interventions: Procedure: Aesthetic Microneedling Treatment
- SkinPen Precision (Active Comparator): Three treatments using SkinPen Precision aesthetic microneedling device to each patient, with each treatment spaced one month apart.
  Interventions: Procedure: Aesthetic Microneedling Treatment

INTERVENTIONS:
Procedure: Aesthetic Microneedling Treatment — Treatment of acne scars on the face and/or back at needle depth settings ranging between 0.25 mm to 2.0 mm, depending on severity and location of scarring.

SUMMARY:
This single-center, clinical trial will take place over a 90 day course followed by 1-month and 6-month post treatment visits to assess the efficacy and tolerability of the SkinPen device when used on both men and women on the face and/or back.

DETAILED DESCRIPTION:
At least 20 subjects of varying Fitzpatrick skin types will be admitted to the trial for treatment on their moderate to severe acne scars on the face and/or back. Implementation of needle depths ranging from 0.25 mm to 2.0 mm will depend on severity of scars and their location. Each subject will undergo 3 treatments in 30 day increments and will take pre-treatment images as well as 1-month and 6-months post treatment images. Assessment will be based on the Goodman and Baron's grading system, the Clinician's Global Aesthetic Improvement Scale, as well as a self-assessment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 60 years of age.
* Subjects in good health.
* Approximately 5 to 10 atrophic acne scars of mixed types (boxcar and/or rolling scars with some icepick scars allowed) on face and/or back that are moderate to severe.
* Desire correction of his/her acne scarring.
* Subjects of child bearing potential must take a urine pregnancy test and must test negative.
* Subjects willing to sign a photography release.
* Willingness to cooperate and participate by following study requirements.

Exclusion Criteria:

* Allergies to facial or general skin care products
* Presence of an active systemic or local skin disease.
* Severe solar elastosis.
* Sensitivity to topical lidocaine.
* Recent history of significant trauma to the face (< 6 months).
* Significant scarring other than acne scars in treated area(s).
* Severe of cystic active and clinically significant acne on the area(s) to be treated.
* History of systemic granulomatous diseases.
* History of hypertrophic or keloid scars.
* Current cancerous or pre-cancerous lesions in area(s) to be treated.
* Had microdermabrasion or glycolic acid treatment to treatment area(s) within 1 month prior to study participation.
* History of chronic drug or alcohol abuse.
* Current smokers or have smoked in the last 5 years.
* History of cosmetic treatments: Skin tightening within last year, injectable filler of any type within the last year, neurotoxins within the last 3 months, ablative resurfacing laser treatments, non-ablative, rejuvanative laser treatments in last 6 months, chemical peel, dermabrasion, non-ablative laser or fractional laser resurfacing of face and neck within the last 4 weeks.
* History of certain prescription medications (accutane or other retinoids, topical retinoids, prescription strength skin lightening devices, anti-wrinkle, skin lightening devices, antiplatelet agents/Anticoagulants, and/or psychiatric drugs).
* Nursing, pregnant, or planning to become pregnant during study.
* Current or pre-existing dermatologic diseases on the face or body (psoriasis, rosacea, eczema, etc.)
* History of immunosupression/immune deficiency disorders.
* Current or history of uncontrolled disease such as asthma, diabetes, hyperthyroidism, etc.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Actual); Study Completion 2017-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Stephens, Ph.D, Principal Investigator — Thomas J. Stephens & Associates, Inc.
Locations (1):
- Stephens & Associates, Richardson, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pre-screening was conducted by phone to determine eligibility criteria through and IRB-approved script. Followed by in-clinic screening visits conducted between December 7, 2015 and February 19, 2016.
Pre-assignment Details: Only participants who met eligibility requirements were enrolled into the study and assigned to groups.
Groups:
- SkinPen II: 21 Subjects, 3 SkinPen II treatments to each patient, each one month apart.
  SkinPen II: Treatment of acne scars on the face and/or back at needle depth settings ranging between 0.25 mm to 2.0 mm, depending on severity and location of scarring.
- SkinPen Precision: 20 Subjects, 3 SkinPen precision treatments to each patient, each one month apart.
  SkinPen Precision: Treatment of acne scars on the face and/or back at needle depth settings ranging between 0.25 mm to 2.0 mm, depending on severity and location of scarring.
Period: Overall Study
Arm/Group | SkinPen II | SkinPen Precision
Started | 21 | 20
Completed | 21 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population includes all participants completing the study.
Groups:
- SkinPen II: 3 treatments with SkinPen II to each patient, each one month apart.
  SkinPen: Treatment of acne scars on the face and/or back at needle depth settings ranging between 0.25 mm to 2.0 mm, depending on severity and location of scarring.
- SkinPen Precision: 3 treatments with SkinPen Precision to each patient, each one month apart.
  SkinPen: Treatment of acne scars on the face and/or back at needle depth settings ranging between 0.25 mm to 2.0 mm, depending on severity and location of scarring.
- Total: Total of all reporting groups
Arm/Group | SkinPen II | SkinPen Precision | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Customized [Mean (Standard Deviation); unit: years] — Men and women 18-60 years of age in generally good health were enrolled after satisfying the inclusion and exclusion criteria. Their age, race, and ethnicity were recorded.
  years
    Completed Subjects | 44.2 (11.4) | 43.8 (12.7) | 44 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Participants were treated and evaluated in Dallas, Texas, USA.
  participants
    United States | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Severity of Acne Scars
Description: Goodman and Baron's Qualitative grading system. Possible scores range from 1 = mild to 4 = severe.
Time Frame: Baseline, 1 month post treatment, and 6 months post treatment
Population: The analysis population includes all participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Skinpen ll: Patients treated with the SkinPen II micro-needling device at 1 day, 30 days and 60 days.
- Skinpen Precision: Patients treated with the SkinPen Precision micro-needling device at 1 day, 30 days and 60 days.
Arm/Group | Skinpen ll | Skinpen Precision
Number analyzed (Participants) | 21 | 20
score on a scale
  Baseline | 3.19 (.40) | 3.10 (.31)
  1-Month Post Treatment | 2.81 (.68) | 2.90 (.55)
  6-Months Post-Treatment | 2.62 (.59) | 2.70 (.57)
Statistical Analysis 1: Comparison: Skinpen ll vs Skinpen Precision; Goodman and Baron's qualitative acne scar severity scores. Calculated from Wilcoxon signed-rank test. Testing hypothesis is that the mean change from baseline is equal to zero; Test type: Superiority; p < 0.008, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Clinician's Global Aesthetic Improvement Assessment (CGAIS)
Description: Clinician's Global Aesthetic Improvement Assessment:
  minimal score is 1- Very much improved and, maximum score is 5 -Worse: The appearance is worse than the original condition
Time Frame: 1 month post treatment, and 6 months post treatment
Population: The analysis population includes all participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skinpen ll | Skinpen Precision
Number analyzed (Participants) | 21 | 20
score on a scale
  1-Month Post Treatment | 3.10 (.77) | 3.20 (.77)
  6-Months Post-Treatment | 2.76 (.77) | 2.70 (.86)
Statistical Analysis 1: Comparison: Skinpen ll vs Skinpen Precision; Null hypothesis 4 (no change); Test type: Superiority; p < .001, Wilcoxen signed-rank test

3. Secondary Outcome: Photo Grading of Acne Scar Assessment
Description: Photo grading of acne scars assessment was done using the following scale [Karnik J. et al, JAAD 2014, 71 (1)]:
  Grade- Term- Description
  0 - Clear-- No depression is seen in the treatment area. Macular discoloration may be seen.
  1. - Very mild- - A single depression is easily noticeable with direct lighting (deep). Most or all of the depressions seen are only readily apparent with tangential lighting (shallow).
  2. - Mild-- A few to several, but less than half of all the depressions are easily noticeable with direct lighting(deep). Most of the depressions see are only readily apparent with tangential lighting (Shallow)
  3- Moderate-- More than half of the depressions are apparent with direct lighting (deep)
  4- Severe-- All or almost all the lesions can be seen with direct lighting (deep)
Time Frame: Day 1 (Baseline), Day 30, Day 60, 1-Month post treatment and 6 Month post treatment
Population: The analyxed population includes all participants who completed the study.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | SkinPen II | SkinPen Precision
Number analyzed (Participants) | 21 | 20
Score on a Scale
  Baseline | 2.81 (0.58) | 2.80 (0.52)
  Day 30 | 2.55 (0.59) | 2.78 (0.57)
  Day 60 | 2.67 (0.53) | 2.70 (0.55)
  1-Month post treatment | 2.71 (0.75) | 2.68 (0.49)
  6-Month post treatment | 2.81 (0.68) | 2.35 (0.59)
Statistical Analysis 1: Comparison: SkinPen II vs SkinPen Precision; Calculated from Wilcoxon signed-rank test. The testing hypothesis is that the mean change from baseline is equal to zero; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Subject Self-Assessment Using SASIS
Description: Subject self-assessment was completed in 2 steps for self-assessed scar improvement scale (SASIS) and subject global aesthetic improvement scale (SGAIS):
  1. Based on a live assessment (subjects were provided with a hand mirror for assessment) of the subject while referring to pre-treatment images.
  2. Based on a comparison of pre-treatment images to current post-treatment images. Rating of Acne Scars
     * 1-Exacerbation of acne scars 0 No change in the appearance of acne scars
       1. 1% - 25% improvement in the appearance of acne scars
       2. 25% - 50% improvement in the appearance of acne scars 3-50% - 75% improvement in the appearance of acne scars 4-75% - 99% improvement in the appearance of acne scars
Time Frame: One Month Post Treatment, 6 Month Post Treatment
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | SkinPen II | SkinPen Precision
Number analyzed (Participants) | 21 | 20
Score on a Scale
  1-Month Post treatment | 1.67 (1.49) | 1.65 (0.93)
  6-Month Post treatment | 1.71 (1.23) | 1.70 (1.08)
Statistical Analysis 1: Comparison: SkinPen II vs SkinPen Precision; Calculated from Wilcoxon signed-rank test. The testing hypothesis is that the mean score is equal to 0 (no change in the appearance of acne scars); Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Subject Self-Assessment Using Global Aesthetic Improvement Scale (SGAIS)
Description: The following rating scale was used for SGAIS:
  Rating and Description
  1. - Very much improved: Optimal cosmetic result
  2. - Much improved: Marked improvement in appearance from the initial condition, but not completely optimal
  3. - Improved: Obvious improvement in appearance from initial condition
  4. -No change: The appearance is essentially the same as the original condition
  5. - Worse: The appearance is worse than the original condition
Time Frame: 1-Month Post Treatment and 6- Month Post Treatment
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- SkinPen Precision: 20 Subjects, 3 SkinPen II treatments to each patient, each one month apart.
  SkinPen Precision: Treatment of acne scars on the face and/or back at needle depth settings ranging between 0.25 mm to 2.0 mm, depending on severity and location of scarring.
Arm/Group | SkinPen II | SkinPen Precision
Number analyzed (Participants) | 21 | 20
Score on a Scale
  1-Month Post Treatment | 2.71 (1.06) | 2.85 (0.75)
  6- Month Post Treatment | 0.91 (1.00) | 2.50 (0.83)
Statistical Analysis 1: Comparison: SkinPen II vs SkinPen Precision; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney); Calculated from Wilcoxon signed-rank test. Testing hypothesis is that the mean score is equal to 4 (no change)

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Description: Adverse Events (AEs) were defined as any untoward medical occurrence regardless of causal relationship with the test article.
Groups:
- SkinPen II: 3 SkinPen ll treatments to each patient, each one month apart.
  SkinPen ll: Treatment of acne scars on the face and/or back at needle depth settings ranging between 0.25 mm to 2.0 mm, depending on severity and location of scarring.
- SkinPen Precision: 3 SkinPen treatments to each patient, each one month apart.
  SkinPen Precision: Treatment of acne scars on the face and/or back at needle depth settings ranging between 0.25 mm to 2.0 mm, depending on severity and location of scarring.
Arm/Group | SkinPen II | SkinPen Precision
All-Cause Mortality (participants affected / at risk) | 0/21 | 1/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 1/21 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SkinPen II (N=21) | SkinPen Precision (N=20)
Anthrapod bite (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Brown recluse - inner right thigh
Erythema (face) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Oedema (face) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (face) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin striae (forehead and both sides of face) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No